CLINICAL TRIAL: NCT06705322
Title: A Phase II, Multicenter Study on the Clinical Effectiveness of Cnidium Monnieri Detoxification Formula for Persistent High-risk Human Papillomavirus Infection of Cervix.
Brief Title: Cnidium Monnieri Detoxification Formula for Persistent High-risk Human Papillomavirus Infection of Cervix.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Libing Xiang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zsfud-HPV-001
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Human Papillomavirus (HPV) Infection; Cervical Cancer
Keywords: Human papillomavirus infection; Cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Cnidium Monnieri Detoxification Formula) (Experimental): Take Cnidium Monnieri Detoxification Formula orally for at least 3 months. Baseline HPV clearance, improvement in clinical symptoms and quality of life, and drug safety were assessed at 3 months, 6 months, and 12 months after initiation of treatment.
  Interventions: Drug: Cnidium Monnieri Detoxification Formula

INTERVENTIONS:
Drug: Cnidium Monnieri Detoxification Formula — Drug composition of Cnidium Monnieri Detoxification Formula: snake seed 9g, Tuckaia 30g, Matrine 9g, snake berry 30g, white Ying 30g. Based on the Cnidium Monnieri Detoxification Formula, the other symptoms were treated with syndrome differentiation and flavor. The traditional Chinese medicine decoction is provided by the Pharmacy of Yueyang Hospital of Integrated Traditional Chinese and Western Medicine Affiliated to Shanghai University of Traditional Chinese Medicine, with 1 dose per day, decocted into 300ml by a medicine decocter, packed in 2 vacuum bags, taken orally after meals, twice a day, one bag each time. Do not stop taking decoction during menstruation. 1 month is a course of treatment, at least 3 courses of treatment, no more than 6 courses of treatment.
  Baseline HPV clearance, improvement in clinical symptoms and quality of life, and drug safety were assessed at 3 months, 6 months, and 12 months after initiation of treatment.

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of Cnidium Monnieri Detoxification Formula in clearing HPV infection, improving clinical symptoms and quality of life in female patients with persistent cervical high-risk HPV infection.

DETAILED DESCRIPTION:
Persistent infection with high-risk HPV is a major cause of cervical cancer and has negative psychosocial effects on women's health-related quality of life (QOL). This prospective, single-arm, multicenter study is to evaluate the clinical efficacy and safety of Cnidium Monnieri Detoxification Formula in clearing HPV infection, improving clinical symptoms and quality of life in female patients with persistent cervical high-risk HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 25 years to ≤ 75 years，with sexual life history
* Meet the diagnostic criteria for high-risk human papillomavirus (HR-HPV) persistent infection
* After surgery or physical therapy for high-grade squamous intraepithelial lesions (HSIL) of the cervix or high-grade squamous intraepithelial lesions (VaINIII) of the vagina, or radical surgery for cervical/vaginal cancer or radical chemoradiotherapy, the examination remained positive for HR-HPV ≥6 months after the end of treatment, with the same type or multiple types as before treatment, and no progression or recurrence of the disease.
* No local or systemic therapy has been administered to patients in the last 3 months
* Patients were informed of the study protocol, agreed to cooperate with the treatment, and signed informed consent.

Exclusion Criteria:

* Only low-risk HPV infection
* Colposcopy for high-grade intraepithelial lesions or cancer of the cervix, vagina, vulva, who have not received or are receiving treatment
* Immunocompromised or immunosuppressant
* Pregnant and lactating women
* Patients with other malignant tumors not controlled, serious heart, lung, liver, renal insufficiency and coagulation dysfunction
* People with communication or cognitive impairment
* Patients have contraindications to oral administration of traditional Chinese medicine preparations
* In the same period, other anti-HPV measures were used to treat, which affected the efficacy judgment

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 79 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-03-27 (Estimated); Study Completion 2027-03-27 (Estimated)

PRIMARY OUTCOMES:
Baseline HPV clearance at 6 months after treatment | 6 months
  HPV clearance rate at 6 months after treatment

SECONDARY OUTCOMES:
Baseline HPV clearance at 12 months after treatment | 12 months
  HPV clearance rate at 12 months after treatment
Safety | 6 months
  Proportion of adverse events within 6 months of treatment

IPD SHARING:
Plan to Share IPD: No